CLINICAL TRIAL: NCT00201994
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Efficacy and Safety Study of the Effects of Titrated Oral Tolvaptan Tablets in Patients With Hyponatremia, Study 2
Brief Title: "SALT-2 Trial" Study of Ascending Levels of Tolvaptan in Hyponatremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Frank Czerwiec, MD PhD, Otsuka Pharmaceutical Development & Commercialization, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-03-238
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Hyponatremia; Water Intoxication; Inappropriate ADH Syndrome; Water-electrolyte Imbalance
Keywords: Sodium; SIADH; Vasopressin; CHF; Cirrhosis; salt; water; electrolyte
MeSH Terms: conditions — Hyponatremia; Water Intoxication; Inappropriate ADH Syndrome; Water-Electrolyte Imbalance; Diabetes Insipidus; Fibrosis | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tolvaptan

SUMMARY:
This study's purpose is to determine whether tolvaptan can safely and effectively return the body's balance of sodium and water toward normal, and to characterize and quantify the potential clinical benefits of this treatment.

DETAILED DESCRIPTION:
Hyponatremia is defined as a serum sodium concentration below the lower limit of normal and is the most frequently encountered electrolyte abnormality in hospitalized patients. Generally speaking, most cases of hyponatremia are mild. However, as the serum sodium falls below 130 mEq/L, the possibility of significant morbidity and mortality increases, and most clinicians will initiate corrective therapy for serum sodium values approaching 130 mEq/L and lower. The reasons for treating hyponatremia relate both to the symptoms, which may be quite disturbing to patients, as well as to potential outcomes including permanent neurological damage and death. there is also growing awareness of the association between hyponatremia and increased mortality in patients with heart failure.

A common theme underlying the occurrence of hyponatremia whether in the setting of congestive heart failure, hepatic failure with ascites, or the syndrome of inappropriate anti-diuretic hormone (SIADH) is the non-osmotic secretion of arginine vasopressin (AVP). The presence of excess AVP leads to fluid retention and hyponatremia. Agents that antagonize AVP, causing proportionally more water diuresis than solute excretion, could offer a significant treatment option for patients with hyponatremia, compared to fluid restriction alone. Treatment of hyponatremia, particularly in clinical settings such as decompensated congestive heart failure, is difficult as conventional diuretics cause neurohormonal activation and further stimulate the inappropriate release of vasopressin, leading to additional retention of free water and aggravation of hypoosmolality. Similarly, for cirrhosis with ascites and SIADH, conventional diuretics are either minimally effective or completely contraindicated. An alternative approach to symptom relief and treatment of hyponatremia may be the use of vasopressin antagonists, which increase free water clearance with proportionally less effect on sodium excretion. Tolvaptan is an oral vasopressin antagonist with relative affinity for the V2 receptor which has been shown to induce a diuresis with proportionally more free-water than sodium loss.

The current study is being undertaken in order to evaluate whether tolvaptan, an oral AVP inhibitor, will be effective in correcting mild to moderate hyponatremia, and to elucidate the effect of this correction on the subject's well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Hyponatremia in euvolemic or hypervolemic states, defined as serum sodium <135 mEq/L prior to randomization.
2. Able to give Informed Consent

Exclusion Criteria:

1. Women who are breast feeding and females of childbearing potential who are not using acceptable contraceptive methods
2. Hyponatremia in hypovolemic states.
3. Acute and transient hyponatremia associated with head trauma or post-operative state.
4. Hyponatremia due to uncontrolled hypothyroidism or uncontrolled adrenal insufficiency.
5. Cardiac surgery within 30 days of potential study enrollment, excluding percutaneous coronary interventions.
6. History of a myocardial infarction within 30 days of potential study enrollment.
7. History of sustained ventricular tachycardia or ventricular fibrillation within 30 days, unless in the presence of an automatic implantable cardioverter defibrillator.
8. Severe angina including angina at rest or at slight exertion and/or unstable angina.
9. History of a cerebrovascular accident within the last 30 days.
10. Subjects with psychogenic polydipsia may not be included, however subjects with other psychiatric illness may be included.
11. Systolic arterial blood pressure <90 mmHg.
12. History of hypersensitivity and/or idiosyncratic reaction to benzazepine or benzazepine derivatives (such as benazepril.).
13. History of drug or medication abuse within the past year,or current alcohol abuse.
14. Uncontrolled diabetes mellitus defined as fasting glucose >300mg/dL.
15. Urinary tract obstruction except BPH if non-obstructive.
16. Previous participation in another clinical drug trial within the past 30 days.
17. Previous participation in this or any other tolvaptan clinical trial.
18. Terminally ill or moribund condition with little chance of short term survival.
19. Serum creatinine >3.5 mg/dL.
20. Serum sodium <120 mEq/L with associated neurologic impairment, i.e. symptoms such as apathy, confusion, seizures.
21. Patients with progressive or episodic neurologic disease such as multiple sclerosis or history of multiple strokes.
22. Child-Pugh score greater than 10 (unless approved)
23. Patients receiving intravenous fluids at a rate greater than KVO (Keep Vein Open).
24. Hyponatremia due to lab artifacts
25. Patients receiving AVP or its analogs for treatment of any condition.
26. Patients receiving within 7 days of randomization, other medications for treatment of hyponatremia specifically: demeclocycline, lithium carbonate or urea
27. Patients likely requiring IV saline for correction of symptomatic or asymptomatic severe hyponatremia during the course of the study.
28. Severe pulmonary artery hypertension
29. Hyponatremia should not be the result of any medication that can safely be withdrawn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2003-11; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The average daily area under the curve of change from baseline in serum sodium level up to Day 4 within the double-blind on therapy period.
and/or
The average daily area under the curve of change from baseline in serum sodium level up to Day 30 within the double-blind on therapy period.

SECONDARY OUTCOMES:
The average daily area under the curve of change from baseline in serum sodium level up to Day 4 within the double-blind on therapy period for patients with severe hyponatremia (serum sodium <130 mEq/L at baseline).
The average daily area under the curve of change from baseline in serum sodium level up to Day 30 within the double-blind on therapy period for patients with severe hyponatremia (serum sodium <130 mEq/L at baseline).
Percentage of patients with normalized serum sodium at Day 4.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Czerwiec, MD, Phd, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (1):
- Universitatskilinikum Carl, Gustav Carus, Dresden, Germany

REFERENCES:
- [Derived] Lee MY, Kang HJ, Park SY, Kim HL, Han E, Lee EK. Cost-effectiveness of tolvaptan for euvolemic or hypervolemic hyponatremia. Clin Ther. 2014 Sep 1;36(9):1183-94. doi: 10.1016/j.clinthera.2014.07.010. Epub 2014 Aug 21. PMID 25151571
- [Derived] Cardenas A, Gines P, Marotta P, Czerwiec F, Oyuang J, Guevara M, Afdhal NH. Tolvaptan, an oral vasopressin antagonist, in the treatment of hyponatremia in cirrhosis. J Hepatol. 2012 Mar;56(3):571-8. doi: 10.1016/j.jhep.2011.08.020. Epub 2011 Oct 23. PMID 22027579
- [Derived] Schrier RW, Gross P, Gheorghiade M, Berl T, Verbalis JG, Czerwiec FS, Orlandi C; SALT Investigators. Tolvaptan, a selective oral vasopressin V2-receptor antagonist, for hyponatremia. N Engl J Med. 2006 Nov 16;355(20):2099-112. doi: 10.1056/NEJMoa065181. Epub 2006 Nov 14. PMID 17105757